CLINICAL TRIAL: NCT06765642
Title: Evaluation of 3 Patterned rTMS Stimulation Dosage on Corticospinal Excitability and Motor Learning in Stroke Patients
Brief Title: The Effect of Non-invasive Brain Stimulation rTMS on Hand Muscles in Chronic Stroke Patients.
Acronym: REALISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00117160
Record Dates: First submitted 2024-12-17; First posted 2025-01-09 (Actual); Last update posted 2025-07-06 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Stroke Patients; Arm Weakness as a Consequence of Stroke; Brain Stimulation; Transcranial Magnetic Stimulation Repetitive; Transcranial Magnetic Stimulation; Motor Learning; Chronic Stroke Patients; Chronic Stroke Survivors
Keywords: stroke; arm weakness; arm weakness as a consequence of stroke; stroke patients; transcranial magnetic stimulation; transcranial magnetic stimulation repetitive; motor learning; chronic stroke; chronic stroke patients; chronic stroke survivors
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Non-invasive Brain Stimulation Modalities (Experimental): All participants will undergo three non-invasive brain stimulation modalities:
  1. Focal conventional iTBS over the ipsilesional motor cortex (i.e., a single bout of 600 pulses over a single spot; FiTBS600).
  2. Focal high dose iTBS over the ipsilesional motor cortex (i.e. 4 bouts of 600 pulses over a single spot = 2400 pulses; FiTBS2400).
  3. Diffuse high dose iTBS over the ipsilesional motor cortex (i.e. 4 bouts of 600 pulses over 4 spots: 600 pulses/spot × 4 spots = 2400 pulses; DiTBS2400)
  Interventions: Diagnostic Test: Transcranial Magnetic Stimulation

INTERVENTIONS:
Diagnostic Test: Transcranial Magnetic Stimulation — The use of this approach aims to potentially maximize motor recovery in chronic stroke by harnessing corticospinal plasticity and modulating motor learning behavior.
  Other Names: Repetitive Transcranial Magnetic Stimulation

SUMMARY:
The study is about using a brain stimulation technique called rTMS (Repetitive Transcranial Magnetic Stimulation) to help improve hand muscles in people who had a stroke. Researchers want to understand how this device can help stroke patients use their hands better.

DETAILED DESCRIPTION:
The goal of this study is to determine the efficacy of a high-dose of a excitatory-specific patterned Transcranial Magnetic Stimulation (i.e., intermittent theta-burst stimulation - iTBS) protocol as a neuromodulatory tool on the neuromotor recovery (corticospinal excitability and motor performance) in individuals with chronic stroke using either the conventional iTBS protocol (600 pulses; iTBS600) or a high dose iTBS protocols (a total of 2400 pulses) over a single spot (Focal iTBS; FiTBS2400) and 4 spots (Diffuse iTBS: DiTBS2400) on the ipsilesional hemisphere. The use of this approach aims to potentially maximize motor recovery in chronic stroke by harnessing corticospinal plasticity and modulating motor learning behavior.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=21 years old of any race or gender
2. First-ever ischemic or hemorrhagic stroke (neuroimaging verified) at least 6 months from stroke onset
3. Unilateral arm weakness measured by FM-UM scale <= 62/64
4. Inducible rest motor threshold and testing motor threshold recorded from the affected first dorsal interosseous (FDI) muscle from the study subject

Exclusion Criteria:

1. Bilateral strokes (infarcts and/or hematoma)
2. Other co-existent neuromuscular disorders affecting upper extremity motor impairment.
3. History of medically uncontrolled depression or other neuropsychiatric disorders despite medications either before or after a stroke that may affect the subject's ability to participate in the study.
4. History of confirmed dementia or taking the following dementia drugs, such as Donepezil, Rivastigmine, Galantamine, Memantine, Aducanumab, Lecanemab, Donanemab that affecting their ability to follow study procedure.
5. Uncontrolled hypertension despite medical treatment(s) at the time of randomization, defined as SBP≥185 mmHg or DBP≥110 mmHg (patient can be treated, reassessed and randomized later).
6. Presence of any MRI/rTMS risk factors including but not limited to:

   1. an electrically, magnetically, or mechanically activated metallic or nonmetallic implant including cardiac pacemaker, intracerebral vascular clips or any other electrically sensitive support system.
   2. a non-fixed metallic part in any part of the body, including a previous metallic injury to the eye.
   3. history of seizure disorder before stroke or seizure after stroke.
   4. preexisting scalp lesion or bone defect or hemicraniectomy.

6. Concurrent enrollment in another interventional stroke recovery study. 7. Concerns that the subject cannot comply with study procedures and visits. 8. Pregnant individuals.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2027-04-13 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
To determine whether there is overall stimulation effect among three stimulation paradigms (FiTBS600; FiTBS2400; DiTBS2400) on the ipsilesional corticospinal excitability of a hand muscle. | Baseline, prior to and after intervention (Pre0 and Pre1; 45 minutes apart)
  Each intervention session (total of 3) will consist of one format of iTBS stimulation. Before and after the intervention, single pulse TMS (spTMS) and motor sequence learning (MSL) will be used to assess the effect of the intervention on corticospinal excitability and motor performance.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Feng, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No